CLINICAL TRIAL: NCT05218421
Title: Carotid Artery Plaque Vulnerability Assessment Using Ultrafast Ultrasound Techniques
Acronym: CAP-VALUE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: Rijnstate Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 112669
Record Dates: First submitted 2022-01-20; First posted 2022-02-01 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Carotid Artery Plaque
Keywords: Ultrasound; Shear wave elastography; Atherosclerotic plaques; Strain elastography; Ultrafast ultrasound flow imaging; Histological plaque characterization
MeSH Terms: conditions — Carotid Stenosis; Plaque, Atherosclerotic | interventions — Ultrasonography, Carotid Arteries; Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Atherosclerotic plaque carotid artery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: Patients with a carotid artery stenosis ≥50% according to clinically performed imaging (i.e. duplex, computed tomography angiography (CTA), or magnetic resonance angiography (MRA)) that are scheduled for a CEA.
  Interventions: Diagnostic Test: Carotid ultrasound; Other: Biospecimen collection and examination; Other: Blood sample collection

INTERVENTIONS:
Diagnostic Test: Carotid ultrasound — Carotid ultrasound with flow and elastography (strain and shear wave) measurements will be performed maximally 2 weeks prior to the CEA. Ultrasound-based flow imaging will be repeated six weeks after the CEA to assess the hemodynamic consequences of the CEA procedure.
Other: Biospecimen collection and examination — The plaque excised during CEA will be histologically examined to assess the plaque composition, and therefore plaque vulnerability.
Other: Blood sample collection — In the first 20 included patients in the Radboudumc, a 10 mL blood sample will be collected during surgery via the arterial line that is applied for regular care.

SUMMARY:
Objective: To explore the association between spatio-temporal blood flow velocities (peak systole and end-diastole at prior-stenosis, at maximum stenosis, and post-stenosis) and carotid plaque vulnerability defined by histology staining. Secondary, to assess the association between ultrasound elastography and carotid plaque vulnerability defined by histology staining. Furthermore, to assess the association between blood flow-derived parameters, including wall shear stress (WSS), vector complexity and vorticity, and plaque vulnerability. To evaluate the hemodynamic consequences of a CEA. Last, to explore whether the presence of circulating biomarkers is related to the degree of plaque vulnerability (as reflected by histology and/or ultrasound).

Study design: A multicentre, prospective, observational, cohort study in a total of 70 patients.

Study population: Patients with a carotid artery stenosis ≥50% according to clinically performed imaging (i.e. duplex, computed tomography angiography (CTA), or magnetic resonance angiography (MRA)) that are scheduled for a CEA.

Intervention (observational): A carotid ultrasound with flow and elastography (strain and shear wave) measurements will be performed maximally 2 weeks prior to the CEA. In the first 20 included patients in the Radboudumc, a 10 mL blood sample will be collected during surgery via the arterial line that is applied for regular care. The plaque excised during CEA will be histologically examined to assess the plaque composition, and therefore plaque vulnerability. Ultrasound-based flow imaging will be repeated six weeks after the CEA to assess the hemodynamic consequences of the CEA procedure. Besides, clinical parameters will be subtracted from electronic health record or, if missing, anamnestically collected from the patient.

Main study parameters/endpoints: Association between 2D spatio-temporal blood flow velocities (peak systole and end-diastole at prior-stenosis, maximum stenosis and post-stenosis), measured by ultrafast ultrasound measurements, and plaque vulnerability (stable versus unstable), defined by histology staining.

ELIGIBILITY:
Inclusion Criteria:

* Presence of carotid artery stenosis (≥50%) according to conventional clinically performed imaging (duplex/CT(A)/MR(A)) and scheduled for a CEA;
* Possibility to perform carotid ultrasound ≤2 weeks before the CEA
* ≥18 years old;
* Able to provide signed or oral informed consent.

Exclusion Criteria:

* Hampered carotid blood flow imaging during clinically performed duplex/doppler measurements due to near to total carotid occlusion at the side of interest or a calcified plaque;
* Restenosis after carotid revascularisation at side of interest;
* Participating in another clinical study, interfering on outcomes;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a carotid artery stenosis ≥50% according to clinically performed imaging (i.e. duplex, computed tomography angiography (CTA), or magnetic resonance angiography (MRA)) that are scheduled for a CEA.
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2022-02-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Assocation between 2D blood flow velocities and plaque vulnerability | Time Frame: max 2 weeks prior to CEA
  Explore the association between 2D spatio-temporal blood flow velocities (peak systole and end-diastole prior-stenosis, at maximum stenosis and post-stenosis) and atherosclerotic carotid plaque vulnerability (stable versus unstable), defined by histology staining.

SECONDARY OUTCOMES:
Association strain and plaque vulnerability | Time Frame: max 2 weeks prior to CEA
  Association between strain parameters and plaque vulnerability (stable versus unstable) quantified by histology staining.
Association shear wave elastography measures and plaque vulnerability | Time Frame: max 2 weeks prior to CEA
  Association between shear wave parameters and plaque vulnerability (stable versus unstable) quantified by histology staining. (only Radboudumc)
Association blood flow-related parameters and plaque vulnerability | Time Frame: max 2 weeks prior to CEA
  Association between blood flow-related parameters, including WSS, vector complexity and vorticity and carotid plaque vulnerability (stable versus unstable) quantified by histology staining.
Comparison predictive value for plaque vulnerability ultrafast imaging techniques vs clinically-used measurements | Time Frame: max 2 weeks prior to CEA
  Comparison between the predictive value for plaque vulnerability (stable versus unstable) of ultrafast imaging techniques (i.e. flow, strain and shear wave elastography) with that of clinically-used duplex measurements.
Status 2D blood flow velocity profiles and flow-related parameters prior- and post-CEA | Time Frame: max 2 weeks prior to CEA and 6 weeks after CEA
  Status of 2D blood flow velocity profiles and flow-related parameters (WSS, vector complexity and vorticity) prior- and post-CEA.
Association circulating inflammatory cytokines and plaque vulnerability | Time Frame: During CEA
  Association between the presence of circulating inflammatory cytokines and the degree of plaque vulnerability (as reflected by histology and/or ultrasound)

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Rijnstate Hospital, Arnhem
  - Radboud university medical center, Nijmegen

IPD SHARING:
Plan to Share IPD: Undecided